CLINICAL TRIAL: NCT04758494
Title: A Study to Assess Quality of Life in Stroke and Multiple Sclerosis Patients of the Same Age Range
Brief Title: Quality of Life Assessment Between Stroke and Multiple Sclerosis Patients of the Same Age Range
Acronym: QoLSMS
Status: Completed | Type: Observational
Sponsor: Hellenic Red Cross Hospital (Other)
Collaborators: G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Roditis, MD, MSc, Chief Resident, Hellenic Red Cross Hospital
Other Study IDs: 257/19-12-2019; 3320/06-02-2020 (Other: Hellenic Red Cross Hospital Administratory Board)
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Multiple Sclerosis; Quality of Life; Depression; Mental Health Disorder
Keywords: stroke; multiple sclerosis; quality of life; mental health; depression; anxiety; well-being; wellness; neurological disorder
MeSH Terms: conditions — Stroke; Multiple Sclerosis; Depression; Mental Disorders; Psychological Well-Being; Anxiety Disorders; Nervous System Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Stroke1-hemiparesis: Patients diagnosed with an ischemic/hemorrhagic stroke and clinical hemiparesis.
  Interventions: Other: Questionnaire
- Stroke 2-mild stroke: Patients diagnosed with an ischemic/hemorrhagic stroke and clinical symptoms of a mild stroke.
  Interventions: Other: Questionnaire
- Stroke 3-speech disorder: Patients diagnosed with an ischemic/hemorrhagic stroke and clinical symptoms of a speech disorder.
  Interventions: Other: Questionnaire
- Stroke 4-hemiparesis mainly of upper limb: Patients diagnosed with an ischemic/hemorrhagic stroke and clinical hemiparesis mainly of upper limb.
  Interventions: Other: Questionnaire
- Stroke 5-memory loss and depression: Patients diagnosed with an ischemic/hemorrhagic stroke and clinical symptoms of memory loss and depression.
  Interventions: Other: Questionnaire
- Multiple Sclerosis: Patients diagnosed with multiple sclerosis.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — In the present study a questionnaire was designed by combining three separate questionnaires, which were weighted for use in Greek population and which are often being used to investigate quality of life of young populations diagnosed with stroke or multiple sclerosis, according to international literature. Those were the following questionnaires: Bathrel (Mahoney et al), Patient Health Questionairre (PHQ-9) (Thomson K et al), Health Survey SF-12 (Kontodinopoulos et al 2007). A draft questionnaire was then created with the addition of questions deemed necessary to provide necessary research information. Overall the questionnaire consisted of 42 questions.
  Part A The first part of the questionnaire included demographics of participants. Part B. The second part of the questionnaire included an assessment of the functionality and independence, an evaluation of experienced depression and an assessment of the quality of life of the target population.

SUMMARY:
The purpose of this study is to investigate the physical, psychological, social and functional aspects of life in relatively young people suffering from vascular stroke and in people diagnosed with multiple sclerosis of the same age group and to generally assess the subjective perception of these patients about their general health and well-being. In addition, to assess the degree of depression experienced by people in this age group who suffer from these diseases. Additional objectives are to investigate important factors that negatively affect the quality of life in this group of patients, according to the international literature, and to highlight targeted interventions to promote mental and physical health in order to improve the quality of life in these chronic patients.

DETAILED DESCRIPTION:
Research on the importance of quality of life in chronic neurological patients has occasionally occupied the international scientific community. Due to the large scale of strokes occurring at young ages as well as multiple sclerosis, more and more research is focusing on the quality of life of these individuals.

The present study is retrospective as well as prospective. The purpose of this study is to investigate the physical, psychological, social and functional aspects of life in relatively young people suffering from vascular stroke and in people diagnosed with multiple sclerosis of the same age group and to generally assess the subjective perception of these patients about their general health and well-being. In addition, to assess the degree of depression experienced by people in this age group who suffer from these diseases. Additional objectives are to investigate important factors that negatively affect the quality of life in this group of patients, according to the international literature, and to highlight targeted interventions to promote mental and physical health in order to improve the quality of life in these chronic patients.

In particular, the research questions that this study is trying to answer are:

* Do young stroke patients exhibit the same quality of life as healthy populations of the same age?
* Do young people with multiple sclerosis have the same quality of life as the healthy population of the same age?
* Do young people with stroke have the same quality of life as patients with multiple sclerosis of the same age?
* Are patients (either with multiple sclerosis or stroke) with almost the same degree of physical independence and are older patients characterized by greater depression and reduced quality of life compared to younger ones?
* Is degree of disability associated with decreased quality of life and increased depression between the two groups of chronic patients?
* Does gender affect the quality of life and the presence of depression?
* Do marital and economic status affect the indicators of depression and quality of life in both populations to be investigated?
* Is location of living a factor that contributes to the reduced quality of life and the triggering of depression in young people with stroke and multiple sclerosis compared to the healthy population?

ELIGIBILITY:
Inclusion Criteria:

* Greek citizenship
* Age 18-60 years
* Hospitalization at the department of Neurology, G. Gennimatas Hospital or at the department of Vascular Surgery and/or Neurosurgery, Hellenic Red Cross Hospital
* Diagnosis of ischemic or hemorrhagic stroke or multiple sclerosis at discharge from hospital

Exclusion Criteria:

* Alien citizenship
* Age below 18 or above 60 years
* Mental or physical disability history before the diagnosis of stroke or multiple sclerosis
* Second stroke during the period of the study
* History of dementia
* Symptoms of aphasia or individuals in comatose state (high NIHS)
* Individuals with stroke in the frontal lobe

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: In the present study the sample were patients with ischemic or hemorrhagic stroke or multiple sclerosis (regardless of EDSS).
  All participants belonged to the age group 18-60, ie they reflected the usual age when the person is professionally active in most parts of the world. These are, after all, the age limits used by the World Health Organization.
  The sample was randomly selected through stratification with representation of patients based on gender, age category and geographical location. Data on age, sex, race, marital status, occupation, educational level, plus morbidity, were identified from medical records and self-reports.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Barthel score | Through study completion, an average of 1 year
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored from 0 (total dependence) up to 3 (total independence), a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL (lowest score=0, highest score=20).
PHQ-9 score | Through study completion, an average of 1 year
  The Patient Health Questionnaire-9 (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The tool rates the frequency of the symptoms which factors into the scoring severity index. Question 9 on the PHQ-9 screens for the presence and duration of suicide ideation. A follow up, non-scored question on the PHQ-9 screens and assigns weight to the degree to which depressive problems have affected the patient's level of function. The PHQ-9 is brief and useful in clinical practice. The PHQ-9 is completed by the patient in minutes and is rapidly scored by the clinician. The higher the total score, the worse the depression the patient exhibits. Minimum score=0 indicates absence of depression, and maximum score=27 indicates severe depression. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
SF12-physical component summary (PCS) score | Through study completion, an average of 1 year
  The Short Form-12 (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. It consists of 12 items, each one scored in a given scale. Each item's scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The physical component of SF-12 measures physical functioning, role limitations due to physical health problems, bodily pain, general health, and vitality (energy/fatigue).
SF12-mental component summary (MCS) score | Through study completion, an average of 1 year
  The Short Form-12 (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. The SF-12 is a shortened version of it's predecessor, the SF-36, which itself evolved from the Medical Outcomes Study. It consists of 12 items, each one scored in a given scale. Each item's scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The mental component of SF-12 measures social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being).
Depression severity level | Through study completion, an average of 1 year
  Depression severity was assessed according to Patient Health Questionnaire-9 (PHQ-9) score from 0-27 (see above) and then characterized by using five distinctive levels, namely: None (0-4), Mild (5-9), Moderate (10-14), Moderate severe (15-19) and Severe (20-27).
Dependency category | Through study completion, an average of 1 year
  Categorization of patient dependency was done according to Barthel score from 0-100 (see above) by using four distinctive categories, namely: Total (0-20), Severe (21-60), Moderate (61-90) and Slight (91-100).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Roditis, MD, MSc, Principal Investigator — Department of Vascular Surgery, Hellenic Red Cross Hospital, Athens, Greece; Theofanis T Papas, MD, MSc, PhD, Study Director — Department of Vascular Surgery, Hellenic Red Cross Hospital, Athens, Greece; Nikolaos Bessias, MD, MSc, PhD, Study Chair — Department of Vascular Surgery, Hellenic Red Cross Hospital, Athens, Greece
Locations (1):
- Department of Vascular Surgery, Hellenic Red Cross Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] WYLIE CM, WHITE BK. A MEASURE OF DISABILITY. Arch Environ Health. 1964 Jun;8:834-9. doi: 10.1080/00039896.1964.10663764. No abstract available. PMID 14157579
- [Background] Imhof L, Suter-Riederer S, Kesselring J. Effects of Mobility-Enhancing Nursing Intervention in Patients with MS and Stroke: Randomised Controlled Trial. Int Sch Res Notices. 2015 Feb 17;2015:785497. doi: 10.1155/2015/785497. eCollection 2015. PMID 27347547
- [Background] Altura KC, Patten SB, Fiest KM, Atta C, Bulloch AG, Jette N. Suicidal ideation in persons with neurological conditions: prevalence, associations and validation of the PHQ-9 for suicidal ideation. Gen Hosp Psychiatry. 2016 Sep-Oct;42:22-6. doi: 10.1016/j.genhosppsych.2016.06.006. Epub 2016 Jul 5. PMID 27638967
- [Background] Hausmann J, Sweeney-Reed CM, Sobieray U, Matzke M, Heinze HJ, Voges J, Buentjen L. Functional electrical stimulation through direct 4-channel nerve stimulation to improve gait in multiple sclerosis: a feasibility study. J Neuroeng Rehabil. 2015 Nov 14;12:100. doi: 10.1186/s12984-015-0096-3. PMID 26577467
- [Background] Yoo SH, Kim SR, So HS, Chung HC, Chae DH, Kim MK, Kim BC, Park MS, Lee SH, Nam TS, Correia H, Cella D. The Validity and Reliability of the Korean Version of the Stigma Scale for Chronic Illness 8-Items (SSCI-8) in Patients with Neurological Disorders. Int J Behav Med. 2017 Apr;24(2):288-293. doi: 10.1007/s12529-016-9593-4. PMID 27900731
- [Background] Thompson K, D'iuso D, Schwartzman D, Dobson KS, Drapeau M. Changes in depressed patients' self-statements. Psychother Res. 2020 Feb;30(2):170-182. doi: 10.1080/10503307.2018.1543976. Epub 2018 Nov 13. PMID 30422103